CLINICAL TRIAL: NCT05083533
Title: Effectiveness of Telerehabilitation on Hamstring Flexibility in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: hazalgenc1
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2021-07

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Evaluation was made before the exercise application, after the eight-week application, and at the sixth month after the exercise program.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tele-rehabilitation (Experimental): For the tele-rehabilitation online group, hamstring stretching exercises were performed with cameras and mutually via online applications.
  Interventions: Behavioral: tele-rehabilitation exercise
- home exercise (Active Comparator): The home exercise group, the exercises were conveyed in the form of a brochure, in written form, on the necessary information. It was recorded how many days the home exercise group did the exercises on a weekly basis.
  Interventions: Behavioral: Home exercise

INTERVENTIONS:
Behavioral: tele-rehabilitation exercise — Telerehabilitation allows patients to interact with providers remotely and can be used both to assess patients and to deliver therapy. Treatment program planned to stretch the muscles of individuals with short hamstring muscle group.
  Stretching exercises for hamstring muscle group shortening were applied 4 days a week, which lasted for 8 weeks in total. For the first four weeks, 3 different stretching exercises per day were planned and performed as 10 seconds of stretching and 5 repetitions. For the last four weeks, 4 different stretching exercises were planned per day and performed with 20 seconds of stretching and 10 repetitions.
  Arms: tele-rehabilitation
Behavioral: Home exercise — All participants received home exercise for 8 weeks. The exercise program includes stretching exercises Stretching exercises for hamstring muscle group shortening were applied 4 days a week, which lasted for 8 weeks in total. For the first four weeks, 3 different stretching exercises per day were planned and performed as 10 seconds of stretching and 5 repetitions. For the last four weeks, 4 different stretching exercises were planned per day and performed with 20 seconds of stretching and 10 repetitions.
  Arms: home exercise

SUMMARY:
the investigators aim is the effectiveness of the tele-rehabilitation exercise program and home exercise program applied to sedentary adults with has shortness of hamstring muscle group

DETAILED DESCRIPTION:
The hamstring muscle group is posterior to the femur and consists of three separate muscles. Biceps femoris long and short head, semitendinosus and semimembranosus.

Hamstring muscle group; proximally, except for the short head of the biceps femoris, the long head of the biceps femoris, semitendinosus and semimembranosus muscles originate from the tuber ischiadicum. Distally, it forms the superolateral (biceps femoris) and superomedial (semimembranosus and semitendinosus) borders of the popliteal fossa. The hamstring muscle group is a biarticular complex that crosses the femoroacetabular and tibiofemoral joints.

The biceps femoris short head is non-biarticular as it originates laterally from the femoral linea aspera distal to the femoroacetabular joint. The main functions of the hamstring muscles are to extend the thigh and flex the knee.

Flexibility is the ability of the joints to move within the range of motion they should be.

Having sufficient flexibility of the hamstring muscle group is an important parameter for an individual to have good body biomechanics and thus a healthy posture in daily life.

Since each individual has a different body biomechanical arrangement, the hamstring muscle group is also of different lengths for each individual. In order to increase the flexibility of a muscle, stretching exercises, which constitute an important part of rehabilitation, are used in the literature and scientific books. Stretching exercises; It is a type of exercise that is frequently preferred in individuals with muscle shortness in order to reduce shortness of muscles, improve flexibility and increase the quality of movement in daily activities of the individual. It is known that the muscle-tendon complex is the structure most affected by stretching exercises. It is stated that this increase in the range of motion of the joint is increased as a result of stretching exercises, and the reason for this increase is due to the characteristics of the static (viscosity and elasticity) and dynamic (neural reflex) components of the connective tissue in the muscle-tendon complex.

While many stretching techniques are used in physiotherapy clinics, static stretching exercises are a frequently used technique due to its ease of application and reliability.

Static stretching exercises; It is the position of lengthening the muscle and holding the muscle at the last tolerable length. Active static stretching exercise is a type of stretching based on voluntary contraction of the antagonist muscle. Studies have shown that active static stretching is more effective in increasing flexibility compared to passive static stretching.

Tele-rehabilitation applications; It is a low-cost, sustainable treatment approach with therapeutic potential the same as standard treatments.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with short hamstring muscle group
* Individuals between the ages of 18-25
* Being a university student

Exclusion Criteria:

* Athletes
* Individuals with orthopedic or neurological problems.
* Surgery history
* Cognitive impairment

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Sit and Reach Test | 5 minutes
  The test was performed with the sit and reach test box, which is used to measure hamstring muscle group shortness. Individuals were asked to sit on a flat surface, put their hands on top of each other with their palms facing the ground, and advance the indicator in the box to the last point they could advance, and perform the test without flexing their knees. The value obtained with Scala C-AAHPERD (Centimeteres) as a result of the measurement of the sit and reach test was recorded in the files of the individuals. Measurements were repeated three times. The averages were calculated and recorded.
Active Straight Leg Raise Test - Goniometer | 5 minutes
  In order to measure the hamstring muscle group shortness, individuals were asked to take the supine position on the bobath bed and raise their legs straight to the last point they could lift. physiotherapists positioned the goniometer on the pivot point, the trochanter major. Individuals were asked to keep their actively raised leg straight and not to cut off the contact of their passive leg from the bed. The goniometric measurement was repeated for both the right and left legs, and the goniometric measurement results were recorded in the files of the individuals. Measurements were repeated three times. The averages were calculated and recorded
Passive Straight Leg Raise Test - Goniometer | 5 minutes
  In order to measure the shortness of the hamstring muscle group, the goniometric measurement was made by passively lifting the leg of the individual in the supine position of the physiotherapist and positioning the goniometer on the trochanter major, which is the pivot point. The goniometric measurement was repeated for both the right and left legs, and the goniometric measurement results were recorded in the files of the individuals. Measurements were repeated three times. The averages were calculated and recorded

SECONDARY OUTCOMES:
International Physical Activity Questionnaire Short Form (IPAQ-SF) | 10 minutes
  The International Physical Activity Questionnaires (IPAQ) comprises a set of 4 questionnaires.
  Long (5 activity domains asked independently) and short (4 generic items) versions for use by either telephone or self-administered methods are available

CONTACTS AND LOCATIONS:
Locations (1):
- Bahçeşehir University, Istanbul, Istanbul Avrupa Kitasi, Turkey (Türkiye)